CLINICAL TRIAL: NCT04070534
Title: Utilization Of A Web-Based Platform (Patient Activated Learning System- PALS) To Improve Knowledge And Follow-Up Among Women With Abnormal Cervical Cancer Screening (PALS)
Brief Title: PALS for Pap Smear Follow up
Acronym: PALS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator is actively pursuing additional funding to continue the work. Once funding is secured, the study will recruit additional patients.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-05020040
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PALS intervention (Other): This arm will influence the development of a patient-directed education module using the Patient Activated Learning System (PALS)
  Interventions: Other: PALS

INTERVENTIONS:
Other: PALS — patient activated learning system

SUMMARY:
In this study, the researchers will utilize information gained from patient interviews about their knowledge of the cervical cancer screening and treatment process, and perceived barriers surrounding appropriate follow up, to create content for the intervention.

DETAILED DESCRIPTION:
The overall goal of this research is to develop and test an intervention designed to improve knowledge and follow up among underserved women with abnormal pap smears. The researchers will use a unique web-based platform, the Patient Activated Learning System (PALS), which provides engaging and informative video and text designed to improve patient knowledge specifically among underserved populations. Twenty diverse patients with abnormal pap smears will be recruited from the Women's Health colposcopy clinic for initial qualitative interviews. Forty patients from the same population will then be engaged in a pre-post pilot to examine feasibility, acceptability, and impact of modules on improving knowledge.

ELIGIBILITY:
Inclusion Criteria:

* All Women 21-65 years with diagnosis of abnormal pap smear presenting to Women's Health Colposcopy Clinic at WCMC
* Access to a smartphone
* English or Spanish Speaking

Exclusion Criteria:

* Pregnant women
* Non-English or Spanish speakers

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reusable knowledge objects (RKOs) | Month 1-2
  Knowledge of cervical cancer screening and treatment, and perceived barriers, as measured in qualitative interviews
Knowledge change | Month 3-4
  Quantitative change in knowledge post-intervention, as measured by attendance rates at follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Eloise Chapman-Davis, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Prebyterian Hospital Weill Cornell, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No